CLINICAL TRIAL: NCT00792584
Title: Patient Preference, Sleep Quality, and Anxiety/Depression: A Randomized Comparison of Etravirine and Efavirenz
Acronym: SWITCH-EE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Bern (Other); University of Lausanne Hospitals (Other); Hospital Lugano (Unknown); University Hospital, Basel, Switzerland (Other); Hospital of Neuchâtel (Unknown)
Responsible Party: Principal Investigator, Alain Nguyen, Dr, Doctor, University Hospital, Geneva
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 08-136
Record Dates: First submitted 2008-11-17; First posted 2008-11-18 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Sleep Disorders
Keywords: etravirine; efavirenz; anxiety; depression; sleep quality; HIV; NNRTI; Tritherapy; compliance; stocrin; To replace efavirenz in long-term users with etravirine; To investigate effect of such replacement on patient preference, sleep quality, daytime sleepiness, and anxiety
MeSH Terms: conditions — Sleep Wake Disorders; Anxiety Disorders; Depression; Sleep Initiation and Maintenance Disorders; Patient Compliance; Disorders of Excessive Somnolence | interventions — etravirine; efavirenz

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): patients treats with etravirine for 6 weeks
  Interventions: Drug: etravirine
- 2 (Experimental): patients treats with efavirenz for 6 weeks
  Interventions: Drug: efavirenz

INTERVENTIONS:
Drug: etravirine — Patient receives etravirine/ placebo or efavirenz / placebo
  Arms: 1
Drug: efavirenz — patient receives efavirenz / placebo or etravirine / placebo
  Arms: 2

SUMMARY:
Efavirenz causes neuropsychiatric side effects and sleep disturbance, including vivid dreams, dizziness, and abnormal tiredness. These symptoms are frequent during the first weeks of treatment, with subsequent attenuation but may not completely resolve even years after efavirenz initiation.

The investigators plan a twelve week, randomized, placebo-controlled, double-blind study. In group 1, efavirenz will be replaced with efavirenz placebo plus etravirine, in group 2, efavirenz would be continued, and etravirine placebo given in addition. After six weeks, patients in group 1 would switch to the regimen of group 2, and vice versa.

The primary endpoint of the trial will be patient preference. Sleep quality, daytime sleepiness, and anxiety will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients > 18 years
* Signing the study consent form and agree to change ART regimen
* Stable HAART including EFV since at least 3 months
* HIV-RNA below 50 copies for at least 3 months

Exclusion Criteria:

* No major psychiatric disease (psychosis, severe depression) diagnosed before the initiation of EFV
* Mentally incompetent patients
* Pregnancy or lactation Women of childbearing potential must use one or two reliable contraceptive methods during the trial, from day 1 to the end of week 12. Acceptable methods include the birth control pill, IUD, condoms with spermicides. Non-acceptable methods include (non-exhaustive list): Withdrawal, calendar (Onigo method), or spermicides alone.
* Concomitant renal or hepatic disease:

  * Creatinine above 150 micromol/L
  * Transaminases above 5 times upper normal limit
  * Prothrombin (Quick) value below 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Symptoms and neurological side effects of study drugs | baseline, week 6 and week 12

SECONDARY OUTCOMES:
Levels of daytime sleepiness | baseline, week 6 and week 12
Sleep Quality | baseline, week 6 and week 12
Patient preference | 12 weeks
Symptoms of depression, anxiety and stress will be assessed | baseline, week 6 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Bernard BH Hirschel, Professor, Principal Investigator — Geneva Hospital
Locations (1):
- Geneva Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- See also: Swiss HIV Cohort Study — http://www.shcs.ch